CLINICAL TRIAL: NCT02769754
Title: Phase III, Randomized, Unblinded, Controlled Clinical Trial for Evaluating the Effectiveness of the Use of the New Hemostatic Patch Hemopatch ® in Patients Undergoing Surgical Liver Resection
Brief Title: Effectiveness of the Use of the New Hemostatic Patch Hemopatch ® in Patients Undergoing Surgical Liver Resection
Acronym: HEMOPATCH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HEMOPATCH
Record Dates: First submitted 2016-05-06; First posted 2016-05-12 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-05

CONDITIONS: Liver Damage; Surgery
Keywords: LIVER; RESECTION; SURGERY

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): In the control group (group A) no additional treatment will be applied after performing the usual surgical hemostasis.
  Interventions: Other: Control
- Hemopatch (Experimental): Hemopatch will be apply in the treatment group (group B), once the standard surgical hemostasis is achieved
  Interventions: Device: Hemopatch

INTERVENTIONS:
Device: Hemopatch — Hemopatch will be apply once the standard surgical hemostasis is achieved.
  Arms: Hemopatch
Other: Control — No additional treatment will be applied after performing the usual surgical hemostasis.
  Arms: Control

SUMMARY:
This prospective randomized study aims to determine the influence of the use of local hemostatic on the incidence of local complications derived from the edge of transection: biliary fistula or bleeding, after scheduled hepatic resection.

DETAILED DESCRIPTION:
Achieving adequate hemostasis is a fundamental prerequisite to successfully perform any surgical procedure, but particularly in cases of visceral abdominal surgery, where a slight bleeding, apparently insignificant, can end in significant bleeding (Haas et al Clinic and Applied thombosis 2006).

Control of intraoperative bleeding is initially performed using traditional techniques such as compression, ligatures, clips, Electrocautery, or clamps. The traditional surgical techniques often fail to prevent bleeding, despite performing a careful and meticulous hemostasis.

The morbidity after elective liver surgery has been reduced in hepatobiliary surgery centers mainly after standardizing anatomical liver resections. These techniques decrease necrosis, bleeding, and the incidence of biliary fistulas (Kraus et al J Am Coll Surg 2005).

Bleeding and biliary fistula are the main determinants of postoperative liver morbidity, with an incidence around 4.2-10% and 4-17% respectively (Yamashita et al Ann Surg 2001; Jin et al World J Gastroenterology 2013).

This complication is difficult to handle especially in patients with cirrhosis or liver cancer, because of reduced platelet and blood coagulation activity (Figueras et al Ann Surg 2007).

Moreover, it is particularly difficult to determine the individual risk of rebleeding or biliary fistula during the intraoperative time.

Many adjuvant surgical hemostatic procedures have been tested in the liver: such as oxidized cellulose, absorbable sponges, fibrillar collagen, and fibrin sealants.

There is an extensive published literature reporting the use of adhesives, Sealants, and topical hemostatics in surgery. There is little doubt that the hemostatic effects of these devices produce a beneficial impact on blood loss. However, there is a wide variation in the literature results. Most of the initial clinical data were obtained in cardiovascular surgery. The only trial that has provided the most significant data in hemostatic efficacy was published by Rousou et al in J Thorac Cardiol South 1999. In this randomized multicenter study, 333 patients that underwent emergency cardiac reoperations were randomized to receive either conventional treatment with fibrinogen or other hemostatic. The 92% of the patients assigned to receive fibrin sealant had a complete hemostasis at 5 minutes, compared with the 12% of those treated with other topical hemostatic.

In clinical practice is difficult to quantify the efficacy of the topical hemostatics on hemostasis. The overall effect of perioperative blood loss can only be inferred indirectly by volume drainage and the number of transfused concentrates (Kraus et al J Am Coll Surg 2005).

The volume of blood loss during liver surgery depends on many factors: systemic coagulation, underlying disease, surgery complexity, surgeon experience, central venous pressure, and local hemodynamics.

Moreover, bile leakages are much harder to identify, define, and particularly to quantify, when compared to bleeding. The biliary system is a low pressure system (less than venous pressure). Animal studies have shown that the use of collagen adhesives is effective for preventing biliary fistulas (Wise et al Am Surg 2002).

In a cohort study of 32 adult patients, in which a right hepatic lobe Split was held, it was compared the use of Tachosil ® versus fibrin glue. The transection area was treated with fibrin glue in 16 patients and with Tachosil ® in the other 16 ones. No differences were observed regarding the need of postoperative transfusion. Nevertheless, the group of patients treated with the fibrin patch showed a significantly lower incidence of bile leakage. Those findings were justified based on the assumption that the use of a fibrin patch, according to its base rich in fibrin, prevents bile leakage, occluding the biliary radicals at the transection (Toti et al Dig Liver Dis. 2010).

The first clinical trial comparing a hemostatic patch (Tachosil ®) versus the standard surgical hemostasis with Argon was published by Frilling et al in 2005 (Frilling et al Langenbecks Arch Surg. 2005). It was observed a reduction in the intraoperative time for hemostasis and less posterior drain in the Tachosil ® group (N = 121).

In 2007, Figueras et al (Figueras et al Ann Surg 2007) published the results of a randomized clinical trial comparing the fibrin glue administration (Tissucol ® + collagen sponge) versus control in 300 patients. The results showed no differences between groups in blood loss, transfusions, and incidence of biliary fistula, and therefore it was concluded that the cessation of the use of fibrin sealant would be a justified saving cost.

In the clinical trial recently published by Moench et al (Langenbecks Arch Surg. 2014) they studied the intraoperative time of hemostasis evaluated at 3 minutes by a non-inferiority design. The collagen hemostatic agent Sangustop ® proved to be as effective as the fibrinogen and thrombin sponge Tachosil ® in times of intraoperative hemostasis (n = 128).

The different results observed among studies may be due to the diversity of the agents evaluated, the poor standardization of the application techniques, and especially by the clinical differences.

Hemopatch® is indicated as a hemostatic device in procedures when the surgical control of bleeding by pressure, ligation, or conventional methods is inefficient or impractical. It consists in a soft, thin, foldable, and flexible collagen patch derived from bovine skin, and NHS-PEG coated (pentaerythritol polyethylene glycol ether tetrasuccinimidil glutarate). The white face, which is applied on the tissue, is covered with a thin layer of NHS-PEG providing a firm adherence to it, thus sealing the bleeding surface and inducing hemostasis at the same time. Because of its flexible structure, the application of Hemopatch ® on the site to achieve hemostasis is easily controlled. The uncoated side is marked with blue squares of a biocompatible dye, to differentiate it from the coated side.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled major or minor liver resection surgery by laparotomy approach.
* Age>18
* They have given their written consent voluntarily after having offered the possibility of their participation in the study.

Exclusion Criteria:

* Pregnancy and lactation
* Patients with urgent surgery
* Concomitant surgery of another organ
* Gallbladder or biliary-enteric anastomosis associated.
* ALPPS surgery (stands for Associating Liver Partition and Portal vein Ligation for Staged hepatectomy).
* Patients with liver transplantation history.
* Patients with previous liver trauma.
* Patients with congenital haematological disease involving clotting factors alteration.
* Patients with known hypersensitivity to bovine proteins and brilliant blue colorante (FD&C Nº1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Bleeding | Day 0 to day 30 (+-10 days)
  Bleeding is defined as the fall of > 3 g/dl of hemoglobin in the postoperative as compared to the baseline value after the operation (the hemoglobin level immediately after surgery) and/or any postoperative transfusion of red blood cells packages because of hemoglobin drop and/or the need for reoperation to stop the bleeding (e.g., embolization or re- laparotomy).
Presence of Biliary Fistula | Day 0 to day 30 (+-10 days)
  Biliary fistula is defined as the presence of high bilirubin levels (Bilirubin> 3x in serum level measured at the same time) in the abdominal drainage, being included the need for interventional radiology due to biliary collection or a re-laparotomy due to biliary fistula (Brooke-Smith et al HPB 2015).

SECONDARY OUTCOMES:
Age | Preoperative
Body Mass Index (BMI) | Preoperative
Gender | Preoperative
Medical history (heart disease, lung disease, cirrhosis) | Preoperative
Hypertension | Preoperative
Dyslipemia | Preoperative
Tobacco | Preoperative
Alcohol | Preoperative
Characteristics of liver disease | Preoperative
  Characteristics of liver disease: benign-malignant (source)
Type of surgery | On surgery
  Type of surgery:Liver resection: major/minor.
Type of surgery | On surgery
  Type of surgery: Number of resected segments/type
Type of surgery | On surgery
  Type of surgery: Number-size of hemostatic patches used as well as their location
Need of transfusion | Day 0 to day 30 (+-10 days)
  concentrates number
Need of transfusion | Day 0 to day 30 (+-10 days)
  blood / plasma / platelet d. intraoperative / postoperative e. blood / plasma / platelet f. concentrates number
Incidence of re-interventions | 30 days after surgery
  Incidence of re-interventions (No / Yes / Number / match)
Postoperative liver failure | Day 5 after surgery
Infection or wound dehiscence | 30 days after surgery
Interventional radiology procedures | 30 days after surgery
  Number of interventional radiology procedures needed and findings
Mortality | 30 days after surgery
  Mortality p.o. (defined as the existence of the event within 30 days p.o.).
Hospital stay (HS) | Up to 30 days after surgery
  Hospital stay (HS) defined as number of days from the preoperative admission to discharge.
Readmissions | From hospital discharge to 30 days after.
  Readmissions (No / Yes / number of days of re-entry / Cause).
Preoperative Chemotherapy Administration | Preoperative
  Up to 30 days after surgery
immunosuppressive therapy | Preoperative
Diuresis | Up to 30 days after surgery
Temperature | Up to 30 days after surgery
Blood preassure | Up to 30 days after surgery
Concomitant medication | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rafael López-Andújar, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robledo AB, Montalva Oron EM, Seller AN, Ibanez JM, Sanz AH, Mizrahi DC, Orbis Castellanos FJ, Andujar RL. Clinical evidence on the use of Hemopatch(R) in reducing bleeding and biliary fistula after liver resection: Prospective randomized study in planned surgery. Cir Esp (Engl Ed). 2025 Dec 17:800270. doi: 10.1016/j.cireng.2025.800270. Online ahead of print. PMID 41418882